CLINICAL TRIAL: NCT00172185
Title: A Study of the Safety and Efficacy of Teduglutide in Subjects With Parenteral Nutrition-Dependent Short Bowel Syndrome Who Completed Protocol CL0600-004 (NCT00081458)
Brief Title: Safety and Efficacy Study of Teduglutide in Subjects With Short Bowel Syndrome Who Completed Protocol CL0600-004 (NCT00081458)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL0600-005; 2004-000439-27 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; Parenteral Nutrition; SBS; Teduglutide
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teduglutide 0.05 mg/kg/d (Experimental): 0.05 mg/kg/d teduglutide subcutaneous injection
  Interventions: Drug: teduglutide 0.05 mg/kg/d
- teduglutide 0.10 mg/kg/d (Experimental): 0.10 mg/kg/d teduglutide subcutaneous injection
  Interventions: Drug: teduglutide 0.10 mg/kg/d

INTERVENTIONS:
Drug: teduglutide 0.05 mg/kg/d — 0.05 mg/kg/d subcutaneous injection
  Other Names: GATTEX
  Arms: teduglutide 0.05 mg/kg/d
Drug: teduglutide 0.10 mg/kg/d — 0.10 mg/kg/d subcutaneous injection
  Other Names: GATTEX
  Arms: teduglutide 0.10 mg/kg/d

SUMMARY:
The purpose of this clinical study is to evaluate the long-term safety and efficacy of daily administration of teduglutide.

DETAILED DESCRIPTION:
Teduglutide is an analog of naturally occurring human glucagon-like peptide-2 (GLP-2), a peptide secreted by L-cells of the distal intestine. GLP-2 is known to increase intestinal and portal blood flow, and inhibit gastric acid secretion. Teduglutide binds to the glucagon-like peptide-2 receptors located in intestinal subpopulations of enteroendocrine cells, subepithelial myofibroblasts and enteric neurons of the submucosal and myenteric plexus. Activation of these receptors results in the local release of multiple mediators including insulin-like growth factor (IGF)-1, nitric oxide and keratinocyte growth factor (KGF).

This multicenter, double-blind, international, Phase III trial will have a treatment period of 28 weeks. Subjects in this study are those who received teduglutide or placebo in protocol CL0600-004 (NCT00081458). These subjects will receive daily subcutaneous injections of 0.05 milligrams or 0.10 milligrams of teduglutide per kilogram of body weight. Subjects will have visits every 4 to 6 weeks and will be assessed for parenteral nutrition (PN) reduction with a follow-up period of 4 weeks duration for those subjects who do not complete this protocol, or do not enter into the long-term safety extension protocol CL0600-010.

ELIGIBILITY:
Inclusion Criteria:

At dosing week 24 of protocol CL0600-004 (NCT00081458), subjects will be reviewed for their participation in this study.

Subjects who meet all of the following criteria can be enrolled in this study:

* Signed and dated informed consent form (ICF) to participate before any study-related procedures are performed
* Completion of protocol CL0600-004 (NCT00081458)

Exclusion Criteria:

* History of cancer or clinically significant lymphoproliferative disease with fewer than 5 years documented disease-free state
* History of alcohol or drug abuse (within previous year)
* Prior use of native glucagon-like peptide 2 (GLP-2) within 3 months of screening visit
* Pregnant or lactating women
* Any condition or circumstance, which in the investigator's opinion would put the subject at any undue risk, prevent completion of the study, or interfere with analysis of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2008-01-24 (Actual); Study Completion 2008-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (21):
- United States (9):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Emory University Hospital, Atlanta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania - Penn Nursing, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
- Hôpital Erasme, Brussels, Belgium
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Hôpital Huriez, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Lariboisière, Paris
- Academic Medical Center, Department of Endocrinology & Metabolism, Amsterdam, Netherlands
- Poland (2):
  - Pracownia Żywienia, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny-Im.prof W.Orłowskiego CMKP, Warsaw
- St. Mark's Hospital, Harrow, United Kingdom

REFERENCES:
- [Result] Jeppesen PB, Gilroy R, Pertkiewicz M, Allard JP, Messing B, O'Keefe SJ. Randomised placebo-controlled trial of teduglutide in reducing parenteral nutrition and/or intravenous fluid requirements in patients with short bowel syndrome. Gut. 2011 Jul;60(7):902-14. doi: 10.1136/gut.2010.218271. Epub 2011 Feb 11. PMID 21317170
- [Result] O'Keefe SJ, Jeppesen PB, Gilroy R, Pertkiewicz M, Allard JP, Messing B. Safety and efficacy of teduglutide after 52 weeks of treatment in patients with short bowel intestinal failure. Clin Gastroenterol Hepatol. 2013 Jul;11(7):815-23.e1-3. doi: 10.1016/j.cgh.2012.12.029. Epub 2013 Jan 17. PMID 23333663
- [Result] Vipperla K, O'Keefe SJ. Study of teduglutide effectiveness in parenteral nutrition-dependent short-bowel syndrome subjects. Expert Rev Gastroenterol Hepatol. 2013 Nov;7(8):683-7. doi: 10.1586/17474124.2013.842894. Epub 2013 Oct 17. PMID 24134154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10Jan2005 - First Subject Enrolled 24Jan2008 - Last Subject Completed
Pre-assignment Details: This was a 28-week study of the safety and efficacy of teduglutide in subjects with parenteral nutrition-dependent short bowel syndrome who completed protocol CL0600-004
Groups:
- Placebo/0.05: Received placebo in Study 004/ Received Teduglutide 0.05 mg/kg/d in Study 005
- Placebo/0.10: Received placebo in Study 004/ Received Teduglutide 0.10 mg/kg/d in Study 005
- 0.05/0.05: Received Teduglutide 0.05 mg/kg/d in Study 004/ Received Teduglutide 0.05 mg/kg/d in Study 005
- 0.10/0.10: Received Teduglutide 0.10 mg/kg/d in Study 004/ Received Teduglutide 0.10 mg/kg/d in Study 005
Period: Overall Study
Arm/Group | Placebo/0.05 | Placebo/0.10 | 0.05/0.05 | 0.10/0.10
Started | 6 | 7 | 25 | 27
Completed | 6 | 5 | 20 | 23
Not Completed | 0 | 2 | 5 | 4
Not completed — Adverse Event | 0 | 1 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — SPONSOR Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/0.05 | Placebo/0.10 | 0.05/0.05 | 0.10/0.10 | Total
Number analyzed (Participants) | 6 | 7 | 25 | 27 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.06) | 56.6 (9.74) | 46.7 (13.48) | 49.4 (14.04) | 48.5 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 10 | 14 | 32
  Male | 2 | 3 | 15 | 13 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 2 | 6
  White | 5 | 7 | 22 | 25 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving a 20% Reduction at Week 28
Description: For those subjects who received teduglutide (0.05 or 0.10 mg dose) in Study 004 and the same in Study 005, Parenteral Nutrition (PN) Use at Week 28 was compared to the Baseline Visit of Study 004 to calculate the 20% reduction in PN Use. For those subjects who received placebo in Study 004 and either teduglutide 0.05 or 0.10 mg dose in Study 005, PN Use at Week 28 was compared to the use of PN at Week 24 of Study 004 to calculate the 20% reduction in PN Use.
Time Frame: 28 weeks
Population: Number of participants for analysis was determined based on completing all of the prerequisite visits in Study 005. Subjects who dropped out of the study were considered failures.
Measure: Number; unit: Participants
Arm/Group | Placebo/0.05 | Placebo/0.10 | 0.05/0.05 | 0.10/0.10
Number analyzed (Participants) | 6 | 7 | 25 | 27
Participants | 5 | 3 | 17 | 14

2. Secondary Outcome: Number of Subjects Who Achieved at Least a One-Day Reduction in Parenteral Nutrition (PN) Use
Description: Number of Subjects Who Achieved at Least a One-Day Reduction in Parenteral Nutrition (PN) Use (Responder Status is Yes or No)
Time Frame: 6 months
Population: Response Status is Yes or No
Measure: Number; unit: participants
Arm/Group | Placebo/0.05 | Placebo/0.10 | 0.05/0.05 | 0.10/0.10
Number analyzed (Participants) | 6 | 7 | 25 | 27
participants
  Response Status: Yes | 4 | 2 | 17 | 10
  Response Status: No | 2 | 5 | 8 | 17

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Treatment-emergent AEs were newly emergent events and/or increased in severity and/or relationship to drug relative to Baseline. AEs prior to Baseline and continued after Randomization were counted only if there was an increase in severity of the event and/or an increase in drug relationship.
Arm/Group | Placebo/0.05 | Placebo/0.10 | 0.05/0.05 | 0.10/0.10
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/7 | 13/25 | 9/27
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 22/25 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo/0.05 (N=6) | Placebo/0.10 (N=7) | 0.05/0.05 (N=25) | 0.10/0.10 (N=27)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GI haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0 (0)
Catheter related complication (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter bacteremia (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 4 (7) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/0.05 (N=6) | Placebo/0.10 (N=7) | 0.05/0.05 (N=25) | 0.10/0.10 (N=27)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (6) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catheter bacteremia (Infections and infestations) | 1 (2) | 1 (3) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 4 (15) | 2 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 4 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (9) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Intestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 2 (3) | 6 (6)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (5) | 2 (2) | 3 (3)
Reproductive system and breast Disorders (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 6 (10)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less